CLINICAL TRIAL: NCT02557984
Title: Dopamine D2/3- and μ-opioid Receptor Antagonists Reduce Cue-induced Reward Responding and Reward Impulsivity in Healthy Volunteers
Brief Title: Dopamine and Opioid Receptor Antagonists Reduce Cue-induced Reward Responding and Reward Impulsivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SNS_Study_01
Record Dates: First submitted 2015-09-14; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Addiction
Keywords: Dopamine; Opioid; Reward
MeSH Terms: conditions — Behavior, Addictive | interventions — Amisulpride; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo Pill
  Interventions: Drug: Placebo
- Amisulpride (Experimental): 400 mg Amisulpride (Solian®)
  Interventions: Drug: Amisulpride
- Naltrexone (Experimental): 50 mg Naltrexone (Naltrexin®)
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Placebo — Placebo Pill
  Other Names: Lactose Placebo Pill
  Arms: Placebo
Drug: Amisulpride — 400 mg Amisulpride
  Other Names: Solian
  Arms: Amisulpride
Drug: Naltrexone — 50 mg Naltrexone
  Other Names: Naltrexin
  Arms: Naltrexone

SUMMARY:
The purpose of this study is to determine how the dopamine and opioid system is involved in reward processing, specifically in cue-induced reward responding and reward impulsivity, using dopamine and opioid receptor antagonists in healthy participants. The investigators predict that particularly the dopamine challenge should alter cue-induced reward responding and reward impulsivity. Such effects would be of high interest for the treatment of disorders which involve impairments of reward processing such as addiction.

DETAILED DESCRIPTION:
In this study the investigators use amisulpride and naltrexone to elucidate what function the dopamine and opioid system have in the processing of reward. Amisulpride [Solian®; sanofi-aventis] is an atypical antipsychotic and acts as an antagonist at dopamine D2 and D3 (D2/D3) receptors with very high specificity. Amisulpride has been used in numerous past studies to study the role of dopamine in the brain, for example in studies on reinforcement learning, memory, and attentional bias in stimulant dependence. Naltrexone [Naltrexin®; OrPha Swiss GmbH] is an opioid antagonist and is clinically used in the management of alcohol and opioid dependence. It has been used to investigate the role of opioid in pain perception, taste detection and recognition, and smoking behavior. The investigators were interested in particular how amisulpride and naltrexone influence cue-induced reward responding and reward impulsivity.

Study Aims

A) Investigating the role of the dopamine system in cue-induced reward responding; B) Investigating the role of the dopamine system in reward impulsivity; C) Investigating the role of the opioid system in cue-induced reward responding; A) Investigating the role of the opioid system in reward impulsivity.

Study Design

This is a double-blind, randomized, placebo-controlled, between-subject blocker study. 121 participants received either placebo, the dopamine D2/D3 receptor antagonist amisulpride (400 mg), or the unselective opioid receptor antagonist naltrexone (50 mg), 3h before the experimental tasks. Subjective effects on mood were assessed by visual analogue scales (VAS). Cue-induced reward responding was measured using a standard Pavlovian-to-Instrumental Transfer (PIT) task, where participants press a button for reward in the presence of a stimulus predicting that reward. Reward impulsivity was measured using a Delay Discounting (DD) Task, in which participants choose between smaller, immediate rewards and larger, delayed rewards.

ELIGIBILITY:
Inclusion Criteria:

* Physically and psychiatrically healthy men and women

Exclusion Criteria:

* Serious past brain disease or injury
* Pacemaker or neurostimulator
* Hearing aid
* Surgery to head or heart
* Potential metal parts in body (metal splinters, gun wounds, shrapnel or surgical clips)
* Neurological or psychiatric problems (including alcoholism, depression, schizophrenia, bipolar disorders, anxiety disorder, claustrophobia, or parkinsonian symptoms)
* High blood pressure, low blood pressure, cardiac attack in anamnesis, irregular heart rate
* Epilepsy
* Emphysema, chest problems, or multiple sclerosis
* Respiratory problems (including difficulty breathing through the nose)
* Pregnancy, nursing, or planning pregnancy
* Diabetes
* Acute Hepatitis
* Allergy or sensitivity to lactose
* Allergy or sensitivity to amisulpride or naltrexone
* Breast cancer or current tumors
* Insufficiency of liver or kidney
* Past use of opiates or other drugs that may interact with amisulpride or naltrexone (such as stimulants)
* Currently taking medications known to interact with amisulpride or naltrexone (including medicines used to treat irregular heart rhythm such as quinidine, disopyramide, amiodarone and sotalol, cisapride, antibiotics such as erythromycin and pentamidine, levodopa, thioridazone (an antipsychotic), or methadone)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cue-Induced Reward Responding Measure | 1 day
  Measured using a Pavlovian-to-Instrumental Transfer Task
Reward Impulsivity Measure | 1 day
  Measured using a Delay Discounting Task

SECONDARY OUTCOMES:
Mood | 1 day
  Current Mood assessed by Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Boris B Quednow, Prof, Principal Investigator — University Hospital of Psychiatry Zurich; Philippe N Tobler, Prof, Principal Investigator — Laboratory for Social and Neural Systems Research, Department of Economics, University of Zurich
Locations (1):
- University Hospital, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Arbisi PA, Billington CJ, Levine AS. The effect of naltrexone on taste detection and recognition threshold. Appetite. 1999 Apr;32(2):241-9. doi: 10.1006/appe.1998.0217. PMID 10097028
- [Background] Gibbs AA, Naudts KH, Spencer EP, David AS. The role of dopamine in attentional and memory biases for emotional information. Am J Psychiatry. 2007 Oct;164(10):1603-9; quiz 1624. doi: 10.1176/appi.ajp.2007.06081241. PMID 17898353
- [Background] Gonzalez JP, Brogden RN. Naltrexone. A review of its pharmacodynamic and pharmacokinetic properties and therapeutic efficacy in the management of opioid dependence. Drugs. 1988 Mar;35(3):192-213. doi: 10.2165/00003495-198835030-00002. PMID 2836152
- [Background] Jocham G, Klein TA, Ullsperger M. Dopamine-mediated reinforcement learning signals in the striatum and ventromedial prefrontal cortex underlie value-based choices. J Neurosci. 2011 Feb 2;31(5):1606-13. doi: 10.1523/JNEUROSCI.3904-10.2011. PMID 21289169
- [Background] Ersche KD, Bullmore ET, Craig KJ, Shabbir SS, Abbott S, Muller U, Ooi C, Suckling J, Barnes A, Sahakian BJ, Merlo-Pich EV, Robbins TW. Influence of compulsivity of drug abuse on dopaminergic modulation of attentional bias in stimulant dependence. Arch Gen Psychiatry. 2010 Jun;67(6):632-44. doi: 10.1001/archgenpsychiatry.2010.60. PMID 20530013
- [Background] Morein-Zamir S, Craig KJ, Ersche KD, Abbott S, Muller U, Fineberg NA, Bullmore ET, Sahakian BJ, Robbins TW. Impaired visuospatial associative memory and attention in obsessive compulsive disorder but no evidence for differential dopaminergic modulation. Psychopharmacology (Berl). 2010 Oct;212(3):357-67. doi: 10.1007/s00213-010-1963-z. Epub 2010 Jul 27. PMID 20661550
- [Background] Rukstalis M, Jepson C, Strasser A, Lynch KG, Perkins K, Patterson F, Lerman C. Naltrexone reduces the relative reinforcing value of nicotine in a cigarette smoking choice paradigm. Psychopharmacology (Berl). 2005 Jun;180(1):41-8. doi: 10.1007/s00213-004-2136-8. Epub 2005 Jan 29. PMID 15682300
- [Background] Lovibond PF, Colagiuri B. Facilitation of voluntary goal-directed action by reward cues. Psychol Sci. 2013 Oct;24(10):2030-7. doi: 10.1177/0956797613484043. Epub 2013 Aug 27. PMID 23982242
- [Derived] Soutschek A, Weber SC, Kahnt T, Quednow BB, Tobler PN. Opioid antagonism modulates wanting-related frontostriatal connectivity. Elife. 2021 Nov 11;10:e71077. doi: 10.7554/eLife.71077. PMID 34761749